CLINICAL TRIAL: NCT04550273
Title: The Effect of Aerobic Exercise on Liver Enzymes in Overweight Prediabetic Patients With Hepatitis c
Brief Title: Leptin and Liver Enzymes Responses to Aerobic Training in Hepatitis c Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: P.T.REC/012/002650
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): The study group (n=20) will receive three sessions of aerobic walking exercise per week for 3 months in addition to the traditional medical treatment
  Interventions: Behavioral: aerobic treadmill exercise
- control group (No Intervention): The control group (n=20) will receive no training

INTERVENTIONS:
Behavioral: aerobic treadmill exercise — The study group (n=20) received three sessions of aerobic exercise per week for 3 months. Every session was done on an electronic treadmill with no inclination started with 5 minutes warm-up then 30 minutes of moderate-intensity aerobic training with 60-75% of target heart rate then followed or ended by 5 minutes cool down.
  Arms: study group

SUMMARY:
Exercise is one of the most vital components of health maintenance. Exercising regularly maintains the cardiovascular system health, promotes the health of liver, and declines the risks of complications induced by CHCV. Since overweight is the main risk factor for IR and type 2 DM which may speed the liver disease progression among HCV patients, exercise is very important for maintenance and loss of weight. Further, exercise can relieve the side effects of medications of HCV, improve immunity, promote a sense of well-being, reduce levels of chronic fatigue, improve blood oxygen levels and increase the endorphins excretion which makes the patients fully energized (Elgendi, Shebl A, Sliem M, and Gary FA, 2018).

Studies on exercise effect in patients with CHCV are quite scarce (de Sousa Fernandes et al., 2019). Decreased leptin levels by exercise positively modulate insulin signaling and inhibit pathology progression (Anaruma et al., 2019). Since studies investigated physical activity effect on regulating HCV related leptin levels are very little, the present study aimed to explore the response of serum leptin and liver enzymes to aerobic exercise in nondiabetic overweight men with CHCV.

DETAILED DESCRIPTION:
The study group (n=20) received three sessions of aerobic walking exercise per week for 3 months. Every session was done on an electronic treadmill with no inclination started with 5 minutes warm-up then 30 minutes of moderate-intensity aerobic training with 60-75% of target heart rate then followed or ended by 5 minutes cool down. The control group (n=20) will receive no training.

ELIGIBILITY:
Inclusion Criteria:

* Men with hepatitis C patients at least from 6 months
* BMI ranged ≥ 25 to < 30 kg/m2.
* fasting blood glucose level (FBG) < 100 mg/dl.
* waist circumference < 102 cm.

Exclusion Criteria:

* Besides the excluded individuals who participated in any form of physical training in the last 6 months, excluded patients by a physician will be patients with acute or other hepatitis types, cirrhotic or hepatocellular carcinoma, renal or respiratory problems, cardiovascular and neurologic diseases, and hypertension

Ages: 40 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — self-representation of gender identity
Enrollment: 40 (Estimated)
Dates: Start 2020-02-09 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Leptin | It will be after 12-week training
  It will be measured in plasma
Liver enzymes | liver enzymes will be after 12-week training
  Serum alanine and aspartate transaminases (AST), (ALT) will be measured in plasma

SECONDARY OUTCOMES:
weight | It will be after 12-week training
  With an empty bladder and stomach, weight will be measured for every participant
Waist circumference (WC) | It will be after 12-week training
  WC will be measured with an inelastic tape at the umbilicus level
fasting blood glucose (FBG) | It will be after 12-week training
  FBG will be measured by On Call ® Plus Acon, REF G113- 214, made in China

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt